CLINICAL TRIAL: NCT00819819
Title: Infant Nutrition and Risk of Celiac Disease: Proposal for an Intervention, Prospective Multicenter Study
Brief Title: Infant Nutrition and Risk of Celiac Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A similar study was conducted and subsequently published in Italy.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Alessio Fasano, Chief of Pediatric Gastroenterology and Nutrition, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2013P000287
Record Dates: First submitted 2009-01-07; First posted 2009-01-09 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Celiac Disease; Infant Nutrition
MeSH Terms: conditions — Celiac Disease | interventions — Glutens; Diet, Gluten-Free

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Gluten containing diet (Active Comparator): Gluten added to diet at 6 months per American Academy of Pediatrics recommendations
  Interventions: Dietary Supplement: Gluten
- 2 Gluten free diet (Active Comparator): Non gluten containing food starch added to diet from 6-12 months
  Interventions: Dietary Supplement: Gluten free diet

INTERVENTIONS:
Dietary Supplement: Gluten — Purified gluten from exaploid wheat introduced per American Academy of Pediatric Recommendations. Three grams from 6-9 months and 5 grams from 9-12 months. The 3-5 grams represents the mean daily intake of gluten during the second half of the first year in infants of different countries.
  Arms: 1 Gluten containing diet
Dietary Supplement: Gluten free diet — Non gluten containing starch added to diet. Three grams from 6-9 months and 5 grams from 9-12 months. After the age of 1 year all children will be allowed age appropriate unrestricted diet.
  Arms: 2 Gluten free diet

SUMMARY:
The study will identify a cohort of infants at risk for celiac disease that can be followed on a long term basis for investigating the natural history the celiac disease based on the pattern of early nutrition. The study will investigate possible early feeding patterns including the timing of introduction to gluten that may protect at least in part from CD development in at risk infants.

DETAILED DESCRIPTION:
From weaning to age 12 months the clinical data, the adherence to the dietary protocol and the amount of intervention baby-food ingested will be checked every month. Following investigations will be performed at the time of recruitment, at time of weaning and at 12, 18, 24, 30,36, 42, 48, 54 and 60 months by taking a sample of blood (maximum 4 ml) from infants (a) quick test for IgA anti-tTG abs determination (few drops); (b) conventional ELISA for serum IgA and IgG anti-tTG determination (0.4 ml);(c) serum zonulin determination (0.1 ml); (e) serum sample for T1D-related autoantibodies (0.25 ml); (f) serum sample to be stocked in the sera bank (0.25 ml); (g) whole blood sample in EDTA for validation of the quick tests (0.5 ml). All the sera samples will be frozen, stored at -20 °C and sent (boxed in dry ice) in blocks to the centre responsible for the determinations every 2 months. Cases positive for the quick-test for anti-tTG the serum sample will be frozen and immediately shipped for confirmatory determination.

If infants develop symptoms during the intervention period (6 to 12 months) the group to which infant belongs will be decoded. Infants belonging to group A (on a gluten-containing diet) presenting symptoms suggestive of CD will undergo a complete diagnostic work-up for CD. These events will be reported in a form. After age 1 year, infants developing symptoms suggestive of active CD (chronic diarrhea, failure to thrive, etc) in-between the scheduled visits will undergo a supplementary serological investigation. A small intestinal biopsy will be recommended in cases showing either serum anti-tTG abs higher than the cut-off or IgG-AGA higher than cut-off in infants with selective IgA deficiency. (Standard medical care and not part of research).

The evolution of the composition of the intestinal microbiota will be evaluated in both groups at 7d, 30d, 4-6 months (prior to weaning), 12,18,24,30,36, 42, 48, 54 and 60 months. The bacterial composition of stool will also be analyzed in a sub-sample of children developing active CD and in non-CD controls. All patients who develop CD will continue in the study.

Definitions:

Active CD: Children showing positive serology and signs of immune-mediated damage of the small intestinal mucosa on biopsy (ranging from isolated increase of intraepithelial lymphocytes to villous atrophy with crypt hypertrophy.)

CD serological autoimmunity positive: Children positive for IgA anti-tTG abs on two consecutive occasions.

Disruption of the small intestinal barrier: Children with an increased ratio of serum lactulose/mannitol with or without increased levels of serum zonulin.

ELIGIBILITY:
Inclusion Criteria:

* Newborns and infants less than 6 months of age
* First-degree relatives of patients affected with biopsy-proven CD
* On exclusive milk diet (breast milk or formula)

Exclusion Criteria:

* Infants that have gluten introduced in their diet before 5-6 months of age
* Infants older than 6 months of age

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2008-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the primary prevention of early onset celiac disease and related autoimmunity phenomena by comparing the frequency of disease development according to two different patterns of gluten introduction in at risk infants | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Alessio Fasano, M.D., Principal Investigator — Center for Celiac Research MGH
Locations (1):
- Massachusetts General Hospital East, Charlestown, Massachusetts, United States

REFERENCES:
- [Background] Ivarsson A, Hernell O, Stenlund H, Persson LA. Breast-feeding protects against celiac disease. Am J Clin Nutr. 2002 May;75(5):914-21. doi: 10.1093/ajcn/75.5.914. PMID 11976167
- [Background] Norris JM, Barriga K, Hoffenberg EJ, Taki I, Miao D, Haas JE, Emery LM, Sokol RJ, Erlich HA, Eisenbarth GS, Rewers M. Risk of celiac disease autoimmunity and timing of gluten introduction in the diet of infants at increased risk of disease. JAMA. 2005 May 18;293(19):2343-51. doi: 10.1001/jama.293.19.2343. PMID 15900004
- [Background] Hoorfar J, Buschard K, Dagnaes-Hansen F. Prophylactic nutritional modification of the incidence of diabetes in autoimmune non-obese diabetic (NOD) mice. Br J Nutr. 1993 Mar;69(2):597-607. doi: 10.1079/bjn19930059. PMID 8490012
- [Background] Norris JM, Barriga K, Klingensmith G, Hoffman M, Eisenbarth GS, Erlich HA, Rewers M. Timing of initial cereal exposure in infancy and risk of islet autoimmunity. JAMA. 2003 Oct 1;290(13):1713-20. doi: 10.1001/jama.290.13.1713. PMID 14519705
- [Background] Funda DP, Kaas A, Bock T, Tlaskalova-Hogenova H, Buschard K. Gluten-free diet prevents diabetes in NOD mice. Diabetes Metab Res Rev. 1999 Sep-Oct;15(5):323-7. doi: 10.1002/(sici)1520-7560(199909/10)15:53.0.co;2-p. PMID 10585617
- [Background] Damci T, Nuhoglu I, Devranoglu G, Osar Z, Demir M, Ilkova H. Increased intestinal permeability as a cause of fluctuating postprandial blood glucose levels in Type 1 diabetic patients. Eur J Clin Invest. 2003 May;33(5):397-401. doi: 10.1046/j.1365-2362.2003.01161.x. PMID 12713453
- [Background] Meddings JB, Jarand J, Urbanski SJ, Hardin J, Gall DG. Increased gastrointestinal permeability is an early lesion in the spontaneously diabetic BB rat. Am J Physiol. 1999 Apr;276(4):G951-7. doi: 10.1152/ajpgi.1999.276.4.G951. PMID 10198339
- [Background] Clemente MG, De Virgiliis S, Kang JS, Macatagney R, Musu MP, Di Pierro MR, Drago S, Congia M, Fasano A. Early effects of gliadin on enterocyte intracellular signalling involved in intestinal barrier function. Gut. 2003 Feb;52(2):218-23. doi: 10.1136/gut.52.2.218. PMID 12524403
- [Background] Watts T, Berti I, Sapone A, Gerarduzzi T, Not T, Zielke R, Fasano A. Role of the intestinal tight junction modulator zonulin in the pathogenesis of type I diabetes in BB diabetic-prone rats. Proc Natl Acad Sci U S A. 2005 Feb 22;102(8):2916-21. doi: 10.1073/pnas.0500178102. Epub 2005 Feb 14. PMID 15710870
- [Background] Sollid LM, Lundin KE. [Disease mechanisms in coeliac disease]. Tidsskr Nor Laegeforen. 2003 Nov 20;123(22):3230-3. Norwegian. PMID 14714017
- [Background] Gronlund MM, Arvilommi H, Kero P, Lehtonen OP, Isolauri E. Importance of intestinal colonisation in the maturation of humoral immunity in early infancy: a prospective follow up study of healthy infants aged 0-6 months. Arch Dis Child Fetal Neonatal Ed. 2000 Nov;83(3):F186-92. doi: 10.1136/fn.83.3.f186. PMID 11040166
- [Background] Kirjavainen PV, Arvola T, Salminen SJ, Isolauri E. Aberrant composition of gut microbiota of allergic infants: a target of bifidobacterial therapy at weaning? Gut. 2002 Jul;51(1):51-5. doi: 10.1136/gut.51.1.51. PMID 12077091
- See also: Related Info — http://www.celiaccenter.org/